CLINICAL TRIAL: NCT00670319
Title: Comparison of Raloxifene Hydrochloride and Placebo in the Treatment of Postmenopausal Women With Osteoporosis
Acronym: MORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1363; H3S-MC-GGGK
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2008-05-01 (Estimated); Status verified 2008-04

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Raloxifene HCL 60 mg orally once a day
  Interventions: Drug: Raloxifene HCL
- 2 (Experimental): Raloxifene HCL 120 mg orally once a day
  Interventions: Drug: Raloxifene HCL
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raloxifene HCL — Raloxifene HCL 60 mg orally once daily
  Other Names: Evista; LY139481
  Arms: 1
Drug: Raloxifene HCL — Raloxifene HCL 120 mg orally once daily
  Other Names: Evista; LY139481
  Arms: 2
Drug: Placebo — Placebo one tab orally per day
  Arms: 3

SUMMARY:
To study the effect of long-term treatment with raloxifene, compared with placebo, on the rate of new vertebral fractures in osteoporotic postmenopausal women with and without existing vertebral fractures.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory postmenopausal women free of severe or chronically disabling conditions, have a life expectancy of at least 5 years, be expected to remain ambulatory throughout the entire study, and be expected to return for follow-up visits.
* Women who have had their last menstrual period at least 2 years before beginning the study.
* Women who have no language barrier, are cooperative, and who give informed consent before entering the study
* Substudy 1:Femoral neck or lumbar spine BMD measurements 2.5 or more standard deviations below normal peak bone mass for healthy, premenopausal women (T-score greater then or equal to 2.5).
* Substudy 2:Either at least one moderate or at least two mild vertebral fractures in the presence of low BMD (as specified above) or at least two moderate vertebral fractures, regardless of BMD.

Exclusion Criteria:

* Patients with known current bone disorders other than primary osteoporosis, such as hyperparathyroidism, Paget's disease, renal osteodystrophy, or osteomalacia
* Patients experiencing clinically severe postmenopausal symptoms at the beginning of the study that require estrogen-replacement therapy
* Patients with known, suspected, or history of carcinoma of the breast or estrogen-dependent neoplasia
* Patients who have had any history of cancer within the previous 5 years
* Patients with abnormal uterine bleeding
* Patients with a history of deep venous thrombosis, thromboembolic disorders, or cerebral vascular accident within the past 10 years except for patients with a history of deep venous thrombosis due to accidents
* Patients who have endocrine disorders requiring pharmacologic therapy except for type II diabetes
* Patients who are not biochemically euthyroid or who have had changes in thyroid replacement therapy in the 2 months before the start of the study.
* Patients with acute or chronic liver disease
* Patients who have impaired kidney function
* Patients with active renal lithiasis
* Patients with known, severe untreated malabsorption syndromes
* Patients with pathologic fractures (both substudies) or patients in Substudy II all of whose vertebral fractures are clearly a result of automobile accidents or other severely traumatic accidents
* Patients in whom satisfactory baseline thoracic and lumbar x-ray views cannot be obtained
* Patients with less than two lumbar and less than four thoracic vertebrae that are unfractured and evaluable for incident fractures
* Treatment with therapeutic doses of any of the following medications more recently than 6 months before beginning the study: Androgen, Calcitonin, Estrogen, Progestin
* Treatment with therapeutic doses of systemic corticosteroids for more than 1 month during the 12 months before beginning the study.
* Patients who have received therapeutic doses of fluorides
* Patients who have received bisphosphonate therapy for more than 14 days during the past 18 months or who have received any bisphosphonate therapy within the last 6 months before beginning the study.
* Patients requiring high-dose heparinization (>7500 U/day) at study entry for a total period of time that will presumably exceed 6 months
* Patients being treated with 50,000 IU or more of vitamin D once weekly more recently than 3 months before beginning the study will be excluded.
* Current systemic treatment with any of the following medications at the beginning of the study: Lithium, Anticonvulsants, regular use of phosphate-binding antacids.

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7705 (Actual)
Dates: Start 1994-11; Primary Completion 1999-09 (Actual); Study Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
To establish the effect of long-term treatment with raloxifene, compared with placebo, on the rate of new vertebral fractures in osteoporotic postmenopausal women with and without prevalent vertebral fractures by spinal x-ray. | Screening, 24, 36, and 72 months
To establish the effect of long-term treatment with raloxifene, compared with placebo, on lumbar spine and femoral neck bone mineral density (BMD) in postmenopausal women with osteoporosis. | Screening, baseline, 12, 24, 36, 48, 60 and 72 months
To establish the safety of chronic administration of raloxifene in postmenopausal women with osteoporosis. Adverse events (AEs), physical exam (PE), EKG, mammograms and laboratory tests will be used to assess safety in the patients. | AEs: throughout the trial. PEs: Randomization, 12, 24, 36, 48, 60, 72 months. ECG: Randomization, 24, 48, 72 months. Mammograms: Randomization, 12, 24, 36, 48, 60, 72 months. Labs: Randomization, baseline, 6, 12, 18, 24, 30, 36, 48, 60, 72 months.

SECONDARY OUTCOMES:
To establish the effect of long-term treatment with raloxifene, compared with placebo, on total body bone mineral content and radial BMD in postmenopausal women with osteoporosis. | Baseline, 24 and 72 months
To establish the effect of raloxifene, compared with placebo, on the rates of new nonvertebral fractures alone & of nonvertebral & vertebral fractures combined in postmenopausal women with osteoporosis by spinal x-ray & assessment of clinical fractures. | Spinal X-rays: Screening, 24, 36 and 72 months. Assessment of clinical fractures: throughout the trial
To establish the effect of long-term treatment with raloxifene, compared with placebo, on biochemical markers of bone metabolism in postmenopausal women with osteoporosis. | Randomization, baseline, 6, 12, 24, 36, and 72 months
To establish the effect of long-term treatment with raloxifene, compared with placebo, on serum lipids and other laboratory markers of cardiovascular risk in postmenopausal women with osteoporosis. | Baseline, 6, 12, 24, 36, and 48 months
To quantify medical resources utilized by patients treated with raloxifene so that a subsequent incremental cost-effectiveness analysis can be performed by quantifying overnight hospitalizations or osteoporotic fractures. | Baseline, 3, 6, 12, 18, 24,30 and 36 months
To assess the impact of raloxifene on quality of life in osteoporotic women with prevalent vertebral fractures by the completion of Quality of Life instruments. | Baseline, 12, 24, and 36 months
To assess the impact of raloxifene on cognitive & neuropsychomotor function using a standardized battery of neuropsychometric tests. | Cognitive/Neuropsychomotor assessments: Baseline, 6, 12, 24, 36, 48, 60 and 72 months
To assess the impact of treatment with raloxifene on risk of cardiovascular disease by monitoring biochemical markers of cardiovascular risk. | Baseline, 6, 12, 24, 36, and 48 months
To assess the possible impact of long-term treatment with raloxifene on risks of endometrial cancer by pelvic gynecological exams and by use of uterine ultrasound in a subset of patients. | GYN Exams and Uterine Ultrasound: Screening, 12, 24, 36, 48, 60 and 72 months.
To assess the possible impact of long-term treatment with raloxifene on breast cancer. | Mammograms: Screening, 24, 36,48 60 and 72 months
To determine the effect of treatment with raloxifene on the prevalence of Alzheimer's disease (AD) on subjects by using a Dementia Diagnostic Evaluation which includes a battery of tests and interviews with the patient as well as brain CT or MRI scan. | Ongoing throughout the trial
To determine the effect of long-term treatment with raloxifene on the prevalence of dementia associated with cerebrovascular (CV) disease in postmenopausal women with osteoporosis by administration of the dementia diagnosis. | Ongoing throughout the trial
Determine the effect of raloxifene on the prevalence of all causes of dementia in subjects by using a Dementia Diagnostic Evaluation which includes a battery of tests and interviews with the patient as well as brain CT or MRI scan. | Ongoing throughout the trial

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad de Buenos Aires, Argentina
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelburg, Australia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz, Austria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels, Belgium
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario, Canada
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague, Czechia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aarhus, Denmark
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turku, Finland
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon, France
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wiesbaden, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest, Hungary
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petach-Tiqva, Israel
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence, Italy
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City, Mexico
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam, Netherlands
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Christchurch, New Zealand
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haugesund, Norway
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok, Poland
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava, Slovakia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ljubljana, Slovenia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona, Spain
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uppsala, Sweden
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London Bridge, United Kingdom

REFERENCES:
- [Derived] Melamed ML, Blackwell T, Neugarten J, Arnsten JH, Ensrud KE, Ishani A, Cummings SR, Silbiger SR. Raloxifene, a selective estrogen receptor modulator, is renoprotective: a post-hoc analysis. Kidney Int. 2011 Jan;79(2):241-9. doi: 10.1038/ki.2010.378. Epub 2010 Oct 6. PMID 20927038